CLINICAL TRIAL: NCT00426049
Title: Monocenter, Double Blinded, Prospective, Randomized Placebo Controlled Study Investigating Prevention of Major Adverse Cardiac Events (MACEs) Within 6 Months by Systemic Treatment With Everolimus After Coronary Intervention With Bare Metal Stents in Patients With Significant Coronary Artery Disease
Brief Title: Systemic Treatment With Everolimus for the Prevention of MACE After Bare Metal Stent Implantation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: German Heart Institute (Other)
Collaborators: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRAD001ADE07
Record Dates: First submitted 2007-01-23; First posted 2007-01-24 (Estimated); Last update posted 2007-01-24 (Estimated); Status verified 2007-01

CONDITIONS: Coronary Artery Disease; Coronary Restenosis
Keywords: Coronary artery disease; Stents; Immunosuppressive Agents; Coronary restenosis; Safety
MeSH Terms: conditions — Coronary Artery Disease; Coronary Restenosis | interventions — Everolimus

INTERVENTIONS:
Drug: Everolimus

SUMMARY:
The purpose of the present study is to provide the first in-human safety and efficacy evaluations of systemic oral anti-proliferative Everolimus therapy compared to placebo in patients treated by bare metal stents for significant coronary artery disease. The aim is to reduce Major Adverse Cardiac Events (MACEs) including death, coronary artery bypass grafting (CABG) to the target vessel, Q-wave and non-Q-wave myocardial infarction, and target lesion revascularization within the first 6 months after intervention. Additionally safety and tolerability of Everolimus at the selected dose in this patient population will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, aged >18 years.
2. Patients with coronary artery disease who are scheduled for coronary intervention with bare metal stent placement for treatment of de novo or first restenosis in a native coronary artery.
3. Target lesion must be in a native coronary vessel of 2.25 - 4.0 mm size.
4. Target lesion has to be of less than or equal to 25 mm length.
5. Tandem lesion may be included as long as:

   * overall length is less than or equal to 25 mm
   * tandem lesion will be treated with one stent and counted as one lesion.

Exclusion Criteria:

The following exclusion criteria must not be present at Baseline visit 1 (BL1, Screening visit prior to coronary intervention). If an exclusion criterion occurred afterwards, e.g., during the coronary intervention, the patient must be excluded from the study.

1. Target lesion has a reference vessel size of less than 2.25 or more than 4.0 mm diameter.
2. Target lesion is a total occlusion or located at a bifurcation.
3. Treatment affords implantation of more than one stent per treated lesion.
4. Target lesion was already treated by brachytherapy.
5. Target lesion has one or more of the following criteria:

   * Left main lesion
   * Ostial lesion of the RCA
   * Located at less than 2 mm after the origin of the LAD or RCX.

Other protocol defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 484
Dates: Start 2006-10

PRIMARY OUTCOMES:
Major adverse cardiac events (MACEs)within 6 months

SECONDARY OUTCOMES:
MACEs within 30 days
Quantitative angiographic observations within the vessel after 6 months
TLR and TVR after 6 months
Drug safety and tolerability for 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Eckart Fleck, Professor, Principal Investigator — German Heart Institute
Locations (1):
- German Heart Institute Berlin, Berlin, State of Berlin, Germany